CLINICAL TRIAL: NCT02334293
Title: Omegaven® as Parenteral Nutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carle Foundation Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13055
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Cholestasis
Keywords: Omegaven; parenteral nutrition; liver disease; liver injury
MeSH Terms: conditions — Cholestasis; Hyperphagia; Liver Diseases | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omegaven (Other)
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — Omegaven® fat emulsion will be used as a Compassionate Use treatment for critically ill infants with PN associated liver injury.

SUMMARY:
The purpose of this study is to determine if a fat emulsion comprised of omega-3 fatty acids, Omegaven, would be beneficial in the management of steatotic liver injury in parenteral nutrition (PN) by its inhibition of de novo lipogenesis, the reduction of arachidonic acid-derived inflammatory mediators, prevention of essential fatty acid deficiency through the presence of small amounts of arachidonic acid, and improved clearance of lipids from the serum.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 14 days old.
* Have PN-associated cholestasis defined as at least 2 consecutive direct bilirubin >2 mg/dL with anatomical or functional short gut (OR >4 mg/dL if intact intestine) obtained at least 1 week apart with a ratio of direct: total bilirubin > 0.4.
* Patients will be PN dependent (unable to meet nutritional needs solely by enteral nutrition) and are expected to require PN for at least 4 more weeks.
* Patients must have failed standard therapies for Parenteral Nutrition Associated Liver Disease (PNALD) including: cycling of PN, avoiding overfeeding, reduction/removal of copper and manganese from PN, advancement of enteral feeding, and use of ursodiol (i.e. Actigall).
* Signed patient informed consent.
* The patient is expected to have a reasonable possibility of survival.
* No other known etiology of cholestasis other than PNALD at time of Omegaven® initiation.

Exclusion Criteria:

* Causes of cholestasis other than PNALD including but not limited to Hepatitis C, Cystic fibrosis, biliary atresia, and alpha 1 anti-trypsin deficiency, prior to Omegaven® initiation.
* Known fish or egg allergy
* Any of the contraindications to use of Omegaven®:

  1. Active new infection at the time of initiation of Omegaven®
  2. Hemodynamic instability
  3. Use of medications with associated risk of bleeding, including nonsteroidal antiinflammatory drugs (NSAIDs)
  4. Active coagulopathy or bleeding
  5. Thrombocytopenia
  6. Unstable hyperglycemia
  7. Impaired lipid metabolism (triglycerides >1000 mg/dL) while on 1 g/kg/day or less of Intralipid
  8. History of severe hemorrhagic disorders (ie. hemophilia, Von Willebrand disease, etc.)
  9. Unstable diabetes mellitus
  10. Collapse and shock
  11. Stroke/ Embolism
  12. Cardiac infarction within the last 3 months
  13. Undefined coma status
* Enrollment in a clinical trial involving an investigational agent (unless approved by the designated physicians on the multidisciplinary team)
* The parent or guardian of child is unwilling to provide consent or assent

Ages: 14 Days to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Primary Outcomes/Endpoints ( time from baseline until the patient normalizes bilirubin (presents three consecutive direct bilirubin ≤ 2 mg/dL or a direct bilirubin ≤ 2 mg/dL and weaned from PN) | Until weaned from PN
  Primary efficacy analysis will include time from baseline until the patient normalizes bilirubin (presents three consecutive direct bilirubin ≤ 2 mg/dL or a direct bilirubin ≤ 2 mg/dL and weaned from PN).

SECONDARY OUTCOMES:
Growth (weight three times per week, length once weekly, and head circumference) | Until weaned from PN
  At a minimum, monitoring of growth parameters while on Omegaven® will include weight three times per week, length once weekly, and head circumference once weekly.
Essential Fatty Acids (evidence of essential fatty acid (EFA) deficiency) | Until weaned from PN
  We will monitor infants who are not receiving any enteral feeding at all for more than 4 weeks for any evidence of essential fatty acid (EFA) deficiency.

CONTACTS AND LOCATIONS:
Overall Officials: William Stratton, MD, Principal Investigator — Carle Foundation Hospital
Locations (1):
- Carle Foundation Hospital, Urbana, Illinois, United States